CLINICAL TRIAL: NCT05343000
Title: A Lifestyle Program for Severe Comorbid Obstructive Sleep Apnea With Severe Obesity
Brief Title: Lifestyle Program for Obstructive Sleep Apnea With Severe Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Minnesota HealthSolutions (Industry)
Responsible Party: Principal Investigator, Roberto P. Benzo, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-011497; R43HL162131 (NIH)
Record Dates: First submitted 2022-04-18; First posted 2022-04-25 (Actual); Results first posted 2025-10-16 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-09

CONDITIONS: Obstructive Sleep Apnea; Obesity
MeSH Terms: conditions — Sleep Apnea, Obstructive; Obesity | interventions — Drug Delivery Systems

STUDY DESIGN:
Intervention Model Description: Pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Severe Comorbid OSA (Experimental): Newly-diagnosed severe comorbid obstructive sleep apnea subjects will use technology to facilitate remote health coaching through a home-based pulmonary rehabilitation (PR) system
  Interventions: Behavioral: Home-based pulmonary rehabilitation (PR) system

INTERVENTIONS:
Behavioral: Home-based pulmonary rehabilitation (PR) system — Technology to facilitate remote health coaching through PAP management, sleep scheduling, sleep duration, diet, exercise, medication and more. The tablet and sensors upload the patient's activities, physiological data, and answers to the daily self-report questions to a secure website. This website also allows health coaches to view patient data via overview, weekly, daily, and trend reports. Health coaches call patients regularly to celebrate progress, assist with any issues, and set new goals.

SUMMARY:
The purpose of this study is to develop a data driven system for persons with severe obesity sleep apnea that utilizes remote monitoring with health coaching to create behavior changes aimed at improving health and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, 18 years of age or older.
* Diagnosis of Obstructive Sleep Apnea (OSA) and obesity (BMI > or = to 35).

Exclusion Criteria:

* Individuals < 18 years of age.
* Patients with an inability to provide good data or follow commands (patients who are disoriented, have a severe neurologic or psychiatric condition).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2024-02-03 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2024-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Benzo, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Severe Comorbid OSA
Started | 17
Completed | 15
Not Completed | 2
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Groups:
- Severe Comorbid OSA: Newly-diagnosed severe comorbid obstructive sleep apnea subjects used technology to facilitate remote health coaching through a home-based pulmonary rehabilitation (PR) system
  Home-based pulmonary rehabilitation (PR) system: Technology to facilitate remote health coaching through PAP management, sleep scheduling, sleep duration, diet, exercise, medication and more. The tablet and sensors uploaded the patient's activities, physiological data, and answers to the daily self-report questions to a secure website. This website also allows health coaches to view patient data via overview, weekly, daily, and trend reports. Health coaches called patients regularly to celebrate progress, assist with any issues, and set new goals.
Arm/Group | Severe Comorbid OSA
Number analyzed (Participants) | 17
Age, Continuous [Mean (Full Range); unit: years] | 54.76 [33 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Ability to Use the Devices at Home
Description: The number of participants who were able to utilize the devices at home.
Time Frame: 2 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Severe Comorbid OSA
Number analyzed (Participants) | 15
Participants | 15

2. Primary Outcome: Usability of Proposed System in Patients With OSA and Obesity
Description: Patients were interviewed by the study coordinator following completion of the intervention. Participants provided feedback on the acceptability and usability of the system, including what they liked and did not like about the interface, the concept of a home-based system, and the health coaching. Participants rated the ease of using the technology on a scale of 1 to 10 (1=very difficult, 10=very easy), with higher scores indicating a better outcome.
Time Frame: 2 Weeks
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Severe Comorbid OSA
Number analyzed (Participants) | 15
score on a scale | 9.5 [1 to 10]

3. Primary Outcome: Helpfulness of Set-up Instructions of Proposed System in Patients With OSA and Obesity
Description: Patients were interviewed by the study coordinator following completion of the intervention. Participants provided feedback on the acceptability and usability of the system, including what they liked and did not like about the interface, the concept of a home-based system, and the health coaching. Participants rated the helpfulness of the setup instructions from 1 to 10 (1=not at all helpful, 10=very helpful), with lower scores indicating a worse outcome.
Time Frame: 2 Weeks
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Severe Comorbid OSA
Number analyzed (Participants) | 15
score on a scale | 9.2 [1 to 10]

4. Secondary Outcome: Participant Reported Confidence Using Proposed System in Patients With OSA and Obesity
Description: Patients were interviewed by the study coordinator following completion of the intervention. Participants provided feedback on the acceptability and usability of the system, including what they liked and did not like about the interface, the concept of a home-based system, and the health coaching. The number of participants who rated their confidence in using the proposed system greater than a 6 on a 10-point scale. The scale ranged from 1=not confident to 10=very confident, with higher scores indicating greater confidence.
Time Frame: 2 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Severe Comorbid OSA
Number analyzed (Participants) | 15
Participants | 15

5. Secondary Outcome: Perceived Benefit of Proposed System in Patients With OSA and Obesity
Description: Patients were interviewed by the study coordinator following completion of the intervention. Participants provided feedback on the acceptability and usability of the system, including what they liked and did not like about the interface, the concept of a home-based system, and the health coaching. The number of participants who rated their perceived benefit from the system greater than a 7 on a 10-point scale. The scale ranged from 1=not beneficial to 10=very beneficial, with higher scores indicating greater benefit.
Time Frame: 2 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Severe Comorbid OSA
Number analyzed (Participants) | 15
Participants | 15

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of informed consent through study completion, approximately 2 weeks.
Arm/Group | Severe Comorbid OSA
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2024-05-24): https://cdn.clinicaltrials.gov/large-docs/00/NCT05343000/Prot_000.pdf